CLINICAL TRIAL: NCT06279026
Title: Single-arm, Open-label, Early-stage Clinical Study of UTAA17 Injection in the Treatment of Relapsed/Refractory Multiple Myeloma
Brief Title: UTAA17 Injection in the Treatment of Relapsed/Refractory Multiple Myeloma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-006-5
Record Dates: First submitted 2024-01-26; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-01

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: UTAA17 injection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UTAA17 Injection (Experimental): After signing informed consent, subjects will be screened according to inclusion/exclusion criteria. Successful subjects will receive 3E8 CAR+γδT, 5E8 CAR+γδT, 1E9 CAR+γδT, 5E9 CAR+γδT, 1E10 CAR+γδT cell transfusions in sequence, and each subject will receive only one dose.
  Interventions: Biological: UTAA17 Injection

INTERVENTIONS:
Biological: UTAA17 Injection — After signing informed consent, subjects will be screened according to inclusion/exclusion criteria. Successful subjects will receive 3E8 CAR+γδT, 5E8 CAR+γδT, 1E9 CAR+γδT, 5E9 CAR+γδT, 1E10 CAR+γδT cell transfusions in sequence, and each subject will receive only one dose.
  Other Names: Chimeric antigen receptor modified T cell injections targeting BCMA

SUMMARY:
The clinical trial was designed as a single-arm, open-label clinical study, with the main purpose of exploring the safety, pharmacokinetics, and best recommended dose (RP2D) of the UTAA17 injection in the treatment of relapsed or refractory multiple myeloma (r/r MM) subjects, and also the efficacy will be observed. Eligible subjects will accept the infusion of UTAA17 injection after pretreatment, and their blood will be collected before and after infusion for evaluation of pharmacokinetics, immunogenicity and safety. This study plans to evaluate efficacy using the revised Evaluation of Efficacy in multiple myeloma -IMWG criteria (2016), which will be evaluated at 4w, 2m, 3m, 6m, and 6 to 24m (at a frequency of Q3m) after cell reinfusion, in addition to the baseline period. Efficacy evaluation continues until one of the following occurs: subject disease progression (PD), acceptance of a new antitumor therapy, death, occurrence of intolerable toxicity, investigator decision, or patient decision to withdraw.

ELIGIBILITY:
Inclusion Criteria:

* All subjects or legal representatives must sign an informed consent form approved by the Ethics Committee in person before commencing any screening process.
* ≥18 years old, regardless of gender, diagnosed with relapsed or refractory multiple myeloma according to the Efficacy Evaluation Criteria for multiple myeloma (IMWG), where relapsed or refractory is defined as: Multiple myeloma that has failed or relapsed after at least 3 lines of therapy (including proteasome inhibitor and immunomodulator-based chemotherapy regimen) in which induction chemotherapy, stem cell transplantation, and maintenance therapy given consecutively are considered a treatment regimen if no disease progression occurs during treatment.
* The presence of measurable lesions at the time of screening will be determined according to any of the following criteria:

  1. Monoclonal plasma cells in bone marrow ≥ 10%.
  2. Serum monoclonal protein (M-protein) level ≥10 g/L.
  3. Urinary M protein level ≥200 mg/24 hours.
  4. Light chain multiple myeloma with no measurable lesions in serum or urine: serum immunoglobulin free light chain ≥10 mg/dL and abnormal serum immunoglobulin κb /γ free light chain ratio.
  5. There are extramedullary lesions.
* BCMA expression on the cell membrane is positive by flow cytometry and/or immunohistochemistry.
* Patients were unable to undergo autologous hematopoietic stem cell transplantation or relapsed after autologous hematopoietic stem cell transplantation and were determined by the investigators to require treatment.
* Patients who have previously received CAR T cell therapy should not be included until at least 3 months after the last CAR T cell infusion and no previously used CAR T cells are detectable in peripheral blood or bone marrow.
* The ECOG score is 0 or 1.
* Expected survival ≥12 weeks.
* Subjects must have appropriate organ function and meet all of the following laboratory test results prior to enrollment

  1. Blood routine: Absolute neutrophil count (ANC) >0.75×10^9 /L; Absolute lymphocyte count (ALC) ≥0.3×10^9 /L; Platelet ≥50×10^9 /L; Hemoglobin >60 g/L
  2. Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × upper limit of normal (ULN); Serum total bilirubin ≤1.5×ULN, except patients with Gilbert syndrome (patients with Gilbert syndrome ≤3.0 times the upper limit of normal and direct bilirubin ≤1.5 times the upper limit of normal can be included)
  3. Renal function: serum creatinine ≤2.5×ULN
  4. Coagulation function: fibrinogen ≥ 1.0g /L; Activated partial thromboplastin time, activated partial thromboplastin time ≤1.5×ULN, and prothrombin time (PT) ≤1.5×ULN
  5. Must have a minimum level of lung reserve, blood oxygen saturation > 92%
* Hemodynamically stable and left ventricular ejection fraction (LVEF) ≥ 50% as determined by echocardiography.

Exclusion Criteria:

* Patients who were determined by the investigators to require long-term immunosuppressant use during screening.
* Cerebrovascular accident or convulsive attack occurred within 6 months before signing the informed consent.
* Other malignancies other than MM, except carcinoma in situ.
* Hepatitis B surface antigen (HBsAg) positive; Hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer detection is not within the normal reference value range; Hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA positive; Human immunodeficiency virus (HIV) antibody positive; cytomegalovirus (CMV) DNA test positive; EBV virus DNA and herpes virus DNA positive test; Syphilis test positive.
* Serious heart disease: including, but not limited to, unstable angina, myocardial infarction (within 6 months prior to screening), congestive heart failure (NYHA classification ≥III), and severe arrhythmia.
* Unstable systemic disease, as determined by the investigator: including, but not limited to, severe liver, kidney, or metabolic disease requiring medical treatment.
* There are chronic progressive neurological disorders.
* Patients who have not yet recovered from the acute toxic effects of prior treatment.
* Presence of active or uncontrolled infections that require systemic treatment (except for mild genitourinary and upper respiratory tract infections).
* Female subjects who are capable of becoming pregnant and plan to become pregnant within 2 years after cell transfusion; Or a male subject whose partner plans to become pregnant within 2 years of cell transfusion.
* The researchers assessed that there were other conditions that were not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
DLT | About 28 days
  Dose limiting toxicity
RP2D | About 1 years
  Best recommended dose

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No